CLINICAL TRIAL: NCT01466335
Title: A Randomized, Double Blind, Parallel Group, Single Center, Adaptive Phase I Study to Evaluate the Safety, Efficacy and Dose Responses of SB-751689 (Ronacaleret; a Calcium Sensing Receptor Antagonist) for Durations Not to Exceed 28 Days, Versusplacebo in Healthy Human Volunteers.
Brief Title: An Adaptive Phase I Study to Evaluate the Safety, Efficacy and Dose Responses of Ronacaleret in Healthy Human Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 115166
Record Dates: First submitted 2011-10-27; First posted 2011-11-07 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Bone Marrow Transplantation
MeSH Terms: interventions — ronacaleret; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Ronacaleret 100mg once daily (Experimental): 1 x 100mg oral tablet
  Interventions: Drug: Ronacaleret (100mg tablet)
- Ronacaleret 100mg twice daily (Experimental): 1 x 100mg oral tablet twice daily
  Interventions: Drug: Ronacaleret (100mg tablet)
- Ronacaleret 200mg once daily (Experimental): 2 x 100mg oral tablet
  Interventions: Drug: Ronacaleret (100mg tablet)
- Ronacaleret 200mg twice daily (Experimental): 2 x 100mg tablets twice daily
  Interventions: Drug: Ronacaleret (100mg tablet)
- Ronacaleret 400mg once daily (Experimental): 4 x 100mg tablets
  Interventions: Drug: Ronacaleret (100mg tablet)
- Placebo (Placebo Comparator): Matching number of identical placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ronacaleret (100mg tablet) — 100mg tablet
  Arms: Ronacaleret 100mg once daily; Ronacaleret 100mg twice daily; Ronacaleret 200mg once daily; Ronacaleret 200mg twice daily; Ronacaleret 400mg once daily
Drug: Placebo — matching placebo tablet
  Arms: Placebo

SUMMARY:
Ronacaleret is an orally administered CaSR antagonist which has previously been demonstrated to transiently increase PTH in both animals and humans. Additional studies in post-menopausal women and patients with distal radial fractures have demonstrated both anabolic and catabolic effects on bone biomarkers and scans of bone density. Based on ronacalerets ability to interact with the CaSR inducing PTH release and activating endogenous bone metabolism of both osteoblasts and osteoclasts, it is our intention to evaluate the impact activation of this pathway has on mobilization of Hematopoietic stem cell (HSCs) into the periphery.

This is an adaptive, phase I, randomized, single centre, double-blind dose finding, parallel-group, multi-cohort placebo controlled study of the efficacy and safety of ronacaleret in up to 45 healthy human volunteers. Cohorts of eligible subjects will be studied for periods up to 28 days. Total daily doses of ronacaleret will range from 100mg, up to 400mg and be administered for a maximum of 28days. The first part of this study will evaluate several doses and schedules of ronacaleret, run in parallel, with respect to their ability to affect mobilization of CD34+ cells into the peripheral circulation. In subsequent cohorts of the study we will utilize information obtained from previous cohorts to further refine and optimise those dosing paradigms which show efficacy. For the first cohort of study participants; the study will commence with 6 days of dosing in an inpatient setting followed by 21 days of continued dosing and evaluation as an outpatient, with a series of regularly scheduled visits, with the final visit on day 28. The study period will include evaluations of pharmacokinetic and pharmacodynamic parameters along with standard laboratory and safety evaluations. The second cohort may be treated with ronacaleret for periods ranging from 14 to 28 days in order to optimise the treatment paradigm with respect to pharmacodynamic efficacy. The PK/PD of each group in cohort one will be utilized to make adjustments in the total daily dose, dose frequency and or duration of dosing investigated in cohort 2. Decisions will be made as to dropping doses based on the PK/PD results and any safety considerations. An initial equal randomization amongst groups within the first cohort may be adjusted to allow for other randomization strategies as various doses and schedules are assessed.

The objective of this study is to characterise the dose-response curve for ronacaleret with respect to safety and efficacy based on changes in peripheral CD34+ cell counts. Results obtained from this study will inform us: of optimized doses, schedules, and durations of treatment for future studies. Additional cohorts may be added to further explore the dose schedule and duration if required. The exact number of cohorts studied will depend on the results obtain from the prior groups and the desire to explore a variety of doses and schedules. The aims of the present study (CR9115166) include an assessment of the pharmacodynamic effects (mobilization of CD34+ cells), safety, tolerability, and pharmacokinetics of ronacaleret in healthy human volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with serum Ca values outside the normal range should always be excluded from enrollment
* Estimated GFR greater than or equal to 60 ml/min/1.73 m2 using the MDRD formula
* AST, ALT, alkaline phosphatase and bilirubin > 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* A female subject is eligible to participate if she is of non-childbearing potential or is of child-bearing potential and agrees to use one of the contraception methods stipulated in the protocol
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol
* Body weight greater than or equal to 55 kg and BMI within the range 20 - 35kg/m2 (inclusive)
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* A positive pre-study HIV, B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of asymptomatic gallstones)
* History of or therapy for osteoporosis
* Subjects taking calcium and/or vitamin D supplements, during or within 2 weeks of study initiation
* Serum calcium (total or albumin-adjusted) outside the central laboratory reference range at the screening visit
* PTH outside the normal range at the screening visit
* Creatine phosphokinase (CPK) outside the normal range at the screening visit
* A positive pre-study drug/alcohol screen
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* Lactating or pregnant females as determined by positive [serum or urine] hCG test at screening or prior to dosing
* Subject is unwilling to refrain from the consumption of red wine, Seville oranges, grapefruit or grapefruit juice [and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices] from 7 days prior to the first dose of study medication until the study visits are complete

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-10-27 (Actual); Primary Completion 2012-03-05 (Actual); Study Completion 2012-03-05 (Actual)

PRIMARY OUTCOMES:
assess the mean fold increase in the number of peripheral CD34+ cells, at total daily doses ranging from 100mg to 400mgs over 1 to 28 days | 1-28 days

SECONDARY OUTCOMES:
Determine the peak CD34+ cell mobilization kinetics | 1-28 days
Adverse Events (AE's) | 1-28 days
optimum dosing frequency respect to mean fold increases in the number of CD34+ cells/kg mobilized | 1-28 days
optimum duration of dosing (ranging from single dose to 28 days) of ronacaleret with respect to mean fold increases in the number of CD34+ cells/kg mobilized | 1-28 days
cardiovascular parameters (12-lead ECG, heart rate, blood pressure) | 1-28 days
clinical chemistry and hematology parameters | 1-28 days
Population pharmacokinetic parameters of GSK962040: Cmax, Tmax, AUC(0-t), Ct, CL/F, V/F, and, if possible, half-life | 1-28 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- See also: Results for study 115166 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115166?search=study&study_ids=115166#rs